CLINICAL TRIAL: NCT03982667
Title: Research Title: Efficacy and Safety of Point- Of-care Procalcitonin Test to Reduce Antibiotic Exposure in Ventilator Associated Pneumonia (VAP) Patient in ICU: A Randomised Controlled Trial
Brief Title: Research Title: Efficacy and Safety of Point- Of-care Procalcitonin Test to Reduce Antibiotic Exposure in VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohd Zulfakar Mazlan, MBBS (Other)
Responsible Party: Sponsor-Investigator, Mohd Zulfakar Mazlan, MBBS, Principle Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: USMalaysia
Record Dates: First submitted 2019-06-08; First posted 2019-06-11 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCT group (Experimental): For patients randomly assigned to the PCT-guided group, measurements of serum PCT concentrations (Day 1, 3, 7, and 9) will be taken and made available to the attending physicians. This means 3 ml of whole blood will be sampled from the arterial line of the patients for each measurement the serum PCT in plain tubes. The samples will be immediately assayed for the PCT measurement using the available device and the results will be ready in next 30 minutes after running the system.
  Interventions: Diagnostic Test: PCT-guided group
- Standard-of-care group (No Intervention)

INTERVENTIONS:
Diagnostic Test: PCT-guided group — In the PCT-guided group, the study protocol encourages to stop the prescribed antibiotics if PCT concentration decrease by 80% or more of its peak value (or if PCT concentration is ≥0·25 and <0·5 μg/L), and strongly encourage to stop the prescribed antibiotics when it reaches a value of < 0·25 μg/L. The attending physician is free to decide whether to continue antibiotic treatment in patients who reach these thresholds. Reasons for non-adherence will be recorded. Antibiotics in the standard-of-care group will be stopped according to local or national guidelines and according to the discretion of attending physicians. Patients will be followed-up until hospital discharge.
  Arms: PCT group

SUMMARY:
Several studies have shown that PCT guidance can reduce the duration of antibiotic treatment for patients with bacterial infections in the ICU, without compromising the safety outcomes. However PCT is known to be more costly than standard biomarkers that commonly use in our ICU setup. This remain the main challenge for us whether by monitoring the PCT level, it can reduce both the duration of antibiotic simultaneously reduce the total cost of the treatment for the patients. A local study addressing efficacy, safety and cost analysis of PCT-guided antibiotic therapy in severe pneumonia patients is therefore warranted. Until the results from a local study become available, the utility of PCT to guide antibiotic duration in our patient population cannot be recommended.

DETAILED DESCRIPTION:
Pneumonia remains one of the major cause of morbidity and mortality in critically ill patients in the intensive care unit (ICU) worldwide. In Malaysia, according to the Malaysian Registry of Intensive Care 2016, pneumonia was among the four (5.7%) most common diagnosis leading to admission to ICU. In many scenario, pneumonia associated with severe sepsis either as single source of sepsis or in combination with other source of infection which carry mortality mortality reported 53.4% 1. Timely, appropriate and adequate antibiotic therapy is of paramount importance in the critically ill patients with severe pneumonia. However, overly long antibiotic treatment is undesirable because of side effects, increasing antibiotic resistance2 and financial burden to patient and Malaysia Healthcare.

Antibiotic remain the main weapon to combat pneumonia. Nevertheless, rampant use of antibiotic without specific indicator is vain. Hence, with the latest technology, physicians not only rely on clinical improvement but also specific biomarkers for resolution of sepsis which might assist the ICU physicians in making decisions on antibiotic therapy on an individual basis.

Commonest used biomarkers for this purpose include leucocyte count and C-reactive protein (CRP). These biomarkers are sensitive but not specific. Procalcitonin (PCT) however has been advocated as a biomarker with a better specificity and sensitivity for diagnosis and follow-up of severe bacterial infections.

PCT is the prohormone of calcitonin. It consists of about 116 amino-acids. The locus of formation in classical pathway is the C-cells of the thyroid. In case of bacterial infection, PCT is formed in all tissues via an alternative pathway. Linscheid et al. 2004 described, in case of bacterial infection two mechanisms of synthesis are at work. At first cytokine-stimulated adherent monocytes release PCT in low quantities. This synthesis is limited. But it plays an important role in the initiation of PCT synthesis in storage tissues of humans. This PCT burst is initiated in all storage tissues (>18h). PCT is a perfect tool to differentiate between viral and bacterial infections (e.g. Gendrel et al. 1999). This is why in septic patients extremely high concentrations of PCT were found in the plasma (about 100,000-fold of the physiological concentration in healthy subjects).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above; and
* Admitted to the ICU; and
* Receive their first dose of antibiotics no longer than 24 h before inclusion to the trial for an assumed or proven bacterial infection.
* Treated as Ventilator Associated Pneumonia (VAP)

Exclusion Criteria:

* Systemic antibiotics as prophylaxis only
* Antibiotics solely as part of selective decontamination of the digestive tract
* Prolonged therapy (eg, endocarditis)
* Expected ICU stay of less than 24 h
* Severe immunosuppression
* Severe infections due to non-bacterial causes
* Previously been enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
To compare the duration of antibiotic treatment between PCT and standard of care groups | 3 to 14 days
  Most of the antiobiotic duration is about 5 - 14 days. In Ventilated Associated Pneumonia, the duration of antibiotic treatment is difficult to stop since the patient stil in intensive care unit due to multiple factors. Therefore the use of PCT guided might be useful.

SECONDARY OUTCOMES:
To compare the mortality between PCT and standard of care | 30 days
  Malaysia Sepsis Mortality rate is nearly 50%. This could be because of higher APACHE score. In PCT guided group, the antibiotic might be stop earlier if clinically indicated. Therefore, the rate of patient die in this group is very important to assess the safety of using this point of care PCT in ICU.
To compare the rate of recurrence infection between PCT and standard of care | 30 days
  By stopping antibiotics earlier, the is possibility risk of recurrent infection if the source of infection is not adequately treated. Therefore the number of recurrence infection is required in PCT group to assess the safety of using PCT guided antibiotic in ICU

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Mohd Zulfakar Mazlan, MBBS, Kota Bharu, Kelantan
  - Mohd Zulfakar Mazlan, Kota Bharu, Kelantan

IPD SHARING:
Plan to Share IPD: No